CLINICAL TRIAL: NCT06043622
Title: Normative Database of Healthy Subject Vascular Density Using Spectralis Heidelberg® Optical Coherence Tomography Angiography
Acronym: COPENBASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: GHPSO de Creil (Unknown); Hôpital Saint Vincent de Paul, Lille (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2023_843_0089
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Optical Coherence Tomography; Optical Coherence Tomography Angiography
Keywords: Normative database; Healthy subjects; Optical coherence tomography; Optical coherence tomography angiography; Heidelberg; Vascular density

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- healthy subject vascular density (Experimental)
  Interventions: Other: Optical coherence tomography angiography; Other: ophthalmological exam

INTERVENTIONS:
Other: Optical coherence tomography angiography — Optical coherence tomography angiography
Other: ophthalmological exam — ophthalmological exam

SUMMARY:
Optical coherence tomography angiography (OCT-A) is a determinant progress to study retinal and choroidal vasculature without using a dye injection. OCT-A yields interesting results in different pathologies such as diabetes mellitus, age-related macular degeneration, hypertension blood pressure, particularly by affecting vascular density. Normative database are necessary to compare OCT-A parameters between patients and controls. However, OCT-A devices from different manufactures may give different values for the same subject. It seems to be obvious that each OCT-A device should have its own normative database. In the literature, OCT-A normative databases are developing using different types of devices, but none is available for Heidelberg OCT-A in Caucasians. The purpose of this project is to create a normative database of retinal microvascularisation using Spectralis Heidelberg optical coherence tomography angiography (OCT-A) ® in normal controls.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary adult subjects or legal representative consenting for minor or subjects under protection
* Intra ocular pression ≤ 21mmHg
* Spherical refraction comprised between - 6 D and +6 D and/or axial length between 21 and 26mm
* Patient affiliated to social security system

Exclusion Criteria:

* Ocular diseases: glaucoma, retinal diseases as diabetic retinopathy, age-related macular degeneration, amblyopia, optic neuropathy
* Diabetes mellitus
* Uncontrolled hypertension blood pressure (> 140/90)
* Recent ocular surgery (< 6 months)
* Any ophthalmological conditions interfering with a good ocular examination or OCT quality (cataract, corneal opacity …)
* OCT-A sufficient quality ≥ 25 (0 = bad quality /40 = excellent quality
* Not consenting patient
* Pathological situation or handicap avoiding good installation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
vascular density of superficial capillary plexus measurement | one day
  vascular density of superficial capillary plexus measurement
vascular density of deep capillary plexus measurement | one day
  vascular density of deep capillary plexus measurement
choriocapillaris density in macular zone | one day
  choriocapillaris density in macular zone
choriocapillaris density in peripapillary zone | one day
  choriocapillaris density in peripapillary zone

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens University Hospital, Amiens, France

IPD SHARING:
Plan to Share IPD: No